CLINICAL TRIAL: NCT01394731
Title: Analgesic Effects of Intravenous Acetaminophen on Labor Pain
Brief Title: Analgesic Effects of Intravenous Paracetamol on Labor Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Collaborators: King Abdulaziz Medical City (Other Government)
Responsible Party: Prof. Jamal A. Alhashemi, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC08-052
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Acetaminophen; Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Paracetamol 1 (Experimental)
  Interventions: Drug: Acetaminophen
- Paraceatmol 2 (Experimental)
  Interventions: Drug: Acetaminophen
- Meperidine (Active Comparator)
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: Acetaminophen
  Arms: Paraceatmol 2; Paracetamol 1
Drug: Meperidine
  Arms: Meperidine

SUMMARY:
The purpose of this study is to determine whether intravenous paracetamol is effective in treating labor pain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I-II
* term patients (≥ 37 weeks of gestation)

Exclusion Criteria:

* previous cesarean section
* hypertension, pre-eclampsia, eclampsia
* intra-uterine growth retardation
* intrauterine fetal death
* morbid obesity (body mass index ≥ 35)
* allergy to any of the study drugs

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score for pain | Up to 24 hours
  Patients who give written informed consent to participate will be entered into the study. Their VAS score will be determined every hour from the time of randomization until delivery of the baby. This time will vary from one patient to another depending on the duration of labor.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Central, Saudi Arabia